CLINICAL TRIAL: NCT04227457
Title: Prospective Epidemiological Study of Metastatic Non Small Cell Lung Cancer (NSCLC) in Latin America
Acronym: LATINO Lung
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0116
Record Dates: First submitted 2018-01-11; First posted 2020-01-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the overall survival of advanced NSCLC in Latin America.

DETAILED DESCRIPTION:
* To describe demographic and socioeconomic characteristics of patients newly diagnosed with advanced NSCLC
* To describe diagnostic methods, pathological profile and disease stage at diagnosis of advanced NSCLC
* To describe the practice patterns of therapeutic agents for treatment of advanced NSCLC
* To describe treatment responses, progression and survival times.
* To describe reasons for treatment discontinuation
* To identify associations between patient demographics, socioeconomic, pathology, treatment sequences and overall survival;
* To define the patient experience of advanced NSCLC and identify unmet needs in their diagnose and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older;
2. Newly diagnosed Non-Small Cell Lung Cancer (NSCLC) during the period of the study (which includes 3 months prior to site activation by LACOG, although they can have received anti-cancer treatment during that time);
3. Histologically or cytologically confirmed advanced NSCLC:

   1. Stage IIIB that progressed after curative therapy (chemoradiation and/or surgery);
   2. Stage IV metastatic disease (de novo or distant relapse)
4. Any NSCLC histological subtype and molecular mutation;
5. Any Eastern Cooperative Oncology Group (ECOG) Performance Status (0 to 4) at diagnosis;
6. Patients assigned by treating physician to any therapy (i.e. chemotherapy, targeted agents, immunotherapy) or palliative care;
7. Access to patient medical chart for data collection;
8. Willing and able to provide written informed consent and privacy authorization for the release of personal health information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The LATINO Lung study will prospectively recruit a minimum of 700 and up to 800 patients with advanced NSCLC, including locally advanced disease not amenable to curative treatment or metastatic disease from sites in Argentina, Brazil, Chile, Colombia, and Mexico. Other countries may be invited to participate.
  Patients will be recruited during an initial study period of 3 months, or more to reach the study minimum sample size, and will be followed for 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Overall survival of advanced NSCLC in Latin America | Annually, during 3 years
  Time from randomization or initiation of treatment to patient death

SECONDARY OUTCOMES:
Description of socioeconomic characteristics of patients newly diagnosed with advanced NSCLC | Annually, during 3 years
  Description of the socioeconomical characteristics of the Latin America population with newly advanced NSCLC
Description of pathological profile of advanced NSCLC | Annually, during 3 years
  Analysis of histology and molecular markers of advanced NSCLC
Description of the practice patterns of therapeutic agents for treatment of advanced NSCLC | Annually, during 3 years
  Description of the practice patterns of therapeutic agents for treatment of advanced NSCLC
Description of the treatment responses | Annually, during 3 years
  Description of the treatment responses
Description of Treatment discontinuation | Annually, during 3 years
  Description of the reasons for treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Barrios, Principal Investigator — Latin American Cooperative Oncology Group; Gustavo Werutsky, Principal Investigator — Latin American Cooperative Oncology Group
Locations (27):
- Argentina (3):
  - Centro Oncologico Riojano, La Rioja, Rioja
  - Instituto De Oncologia De Rosario, Santa Fe, Rosário
  - Centro Medico San Roque, Córdoba, Tucumán Province
- Brazil (18):
  - CRIO, Fortaleza, Ceará
  - CLION, Salvador, Estado de Bahia
  - NOB, Salvador, Estado de Bahia
  - Hospital Sírio- Libanês, Brasília, Federal District
  - ICTr, Curitiba, Paraná
  - Hospital de Câncer de Londrina, Londrina, Paraná
  - Hospital de Caridade de Carazinho, Carazinho, Rio Grande do Sul
  - CPO, Porto Alegre, Rio Grande do Sul
  - HCPA, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Clínica Reichow, Blumenau, Santa Catarina
  - CNT Itajaí, Itajaí, Santa Catarina
  - Barretos, Barretos, São Paulo
  - COI Américas, Rio de Janeiro
  - INCA, Rio de Janeiro
  - AC Camargo, São Paulo
  - IBCC, São Paulo
- Fundación Arturo López Pérez, Providencia, Santiago Metropolitan, Chile
- Colombia (3):
  - Clínica del Country, Chapinero, Bogota D.C.
  - Oncomedica, Montería, Departamento de Córdoba
  - Hospital Pablo Tobon Uribe, Robledo, Medellín
- Mexico (2):
  - Centro Médico Nacional Siglo XXI, Mexico City, Not Aplicable
  - INCan, Mexico City, Not Aplicable

IPD SHARING:
Plan to Share IPD: Undecided